CLINICAL TRIAL: NCT07214142
Title: Efficacy and Safety of Total Neoadjuvant Chemoradiotherapy Combined With PD-1 Therapy for Locally Advanced Rectal Cancer With High Risk of Recurrence
Brief Title: Total Neoadjuvant Therapy With PD-1 for Locally Advcancer Rectal Cancer
Acronym: TNT-Immunity
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Principal Investigator, Liu Liu, Principal Investigator, The First Affiliated Hospital of University of Science and Technology of China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FirstAHUSTCina
Record Dates: First submitted 2025-09-25; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Rectal Cancer Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TNT-immunity (Experimental): 1
  Interventions: Drug: PD-1

INTERVENTIONS:
Drug: PD-1 — patients will receive short-course chemotherapy and concurrent PD-1

SUMMARY:
Research Objective:To investigate the efficacy and safety of the "total neoadjuvant chemoradiotherapy combined with immunotherapy" regimen for the treatment of locally advanced rectal cancer with high-risk features for recurrence.

Study Design:A single-arm, multicenter clinical study.

Study Population: Patients with locally advanced rectal cancer presenting with high-risk features for local recurrence.

DETAILED DESCRIPTION:
Study Title:A Single-Arm, Multicenter Clinical Study to Evaluate the Efficacy and Safety of Total Neoadjuvant Chemoradiotherapy Combined with PD-1 Inhibitor Immunotherapy in Locally Advanced Rectal Cancer with High-Risk Features for Recurrence

Background and Rationale:

Locally advanced rectal cancer (LARC) with high-risk features, such as involved mesorectal fascia, extramural vascular invasion, or low-lying tumors, is associated with a significant risk of local recurrence and distant metastasis following standard treatment. Total neoadjuvant therapy (TNT), which administers both chemotherapy and chemoradiotherapy prior to surgery, has emerged as a strategy to improve pathological outcomes and systemic control. The integration of immune checkpoint inhibitors, specifically PD-1 inhibitors, into TNT regimens is a promising approach. It is hypothesized that radiotherapy may potentiate the immune response by increasing tumor antigen exposure, thereby enhancing the efficacy of immunotherapy and potentially leading to higher rates of complete response and improved long-term survival.

Primary Objective:

The primary objective of this study is to evaluate the efficacy of the combined TNT and PD-1 inhibitor regimen, as measured by the pathological complete response (pCR) rate, defined as the absence of viable tumor cells in the primary tumor and lymph nodes upon pathological examination after surgical resection.

Secondary Objectives:

Secondary objectives are to further assess the treatment's efficacy and safety, including:

Rate of Clinical Complete Response (cCR):The proportion of patients achieving a complete response based on clinical, endoscopic, and radiological assessments prior to surgery.

R0 Resection Rate:The proportion of patients undergoing surgery with microscopically negative margins.

Tumor Regression Grade (TRG):The degree of tumor cell destruction scored by pathological assessment.

Event-Free Survival (EFS):The time from treatment initiation to disease progression, recurrence, or death from any cause.

Overall Survival (OS):The time from treatment initiation to death from any cause.

Safety and Tolerability:The incidence and severity of adverse events, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), with a specific focus on immune-related adverse events (irAEs).

Study Design:

This is a single-arm, open-label, multicenter, Phase II clinical study**. All enrolled participants will receive the same investigational treatment regimen.

Study Population:

The study will enroll adult patients (age ≥ 18 years) with histologically confirmed, locally advanced rectal adenocarcinoma. Eligible participants must have high-risk features for recurrence, which may include:

Clinical stage T3-4 and/or N2 disease. Threatened or involved mesorectal fascia (MRF+). Presence of extramural vascular invasion (EMVI+). Low-lying tumors where sphincter preservation is a concern. Patients must have an ECOG performance status of 0-1 and adequate organ function.

Intervention:

Patients will receive the "Total Neoadjuvant Chemoradiotherapy Combined with Immunotherapy" regimen, which consists of:

1. Induction Immunochemotherapy:Combination of a PD-1 inhibitor (e.g., Pembrolizumab or Nivolumab) with CAPOX or FOLFOX chemotherapy for a specified number of cycles.
2. Chemoradiotherapy:** Concurrent administration of radiotherapy (total dose of 25 Gy in 5 fractions) with a radiosensitizing fluoropyrimidine chemotherapy (e.g., capecitabine).
3. Consolidation Immunotherapy:Additional cycles of the PD-1 inhibitor following chemoradiation.

Surgical resection (Total Mesorectal Excision) will be performed approximately 8-12 weeks after the completion of all neoadjuvant therapy.

Statistical Analysis:

The pCR rate will be summarized with a 95% confidence interval. Secondary time-to-event endpoints like EFS and OS will be estimated using the Kaplan-Meier method. Safety analysis will include all patients who received at least one dose of the study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed rectal adenocarcinoma;
2. Mid-low rectal cancer, with the lower edge of the tumor located within 12 cm from the anal verge;
3. Magnetic resonance imaging (MRI) suggests locally advanced rectal cancer (T3 or T4 and M0), accompanied by at least one of the following risk factors: cT4, N2, lymphovascular invasion, involvement of the mesorectal fascia, or enlarged lateral lymph nodes (short-axis diameter > 8 mm); patients with potentially resectable disease;
4. Polymerase chain reaction (PCR) testing indicates microsatellite stability (MSS) type;
5. No prior antitumor therapy, such as chemotherapy, radiotherapy, immunotherapy, or targeted therapy;
6. Age between 18 and 75 years;
7. ECOG Performance Status (PS) score of 0-1;
8. Laboratory test results: WBC ≥ 3.5 × 10^9/L, Hb ≥ 100 g/L, PLT ≥ 100 × 10^9/L; normal liver and kidney function;
9. Absence of severe comorbidities, and ability to tolerate surgical treatment;
10. The patient or their immediate family member voluntarily agrees to participate in this study and provides written informed consent.

Exclusion Criteria:

1. Recurrent rectal cancer;
2. Synchronous colorectal cancer;
3. Pregnant or lactating patients;
4. History of other malignant tumors;
5. Previous antitumor therapy, including chemotherapy or radiotherapy;
6. Dysfunction of vital organs such as cardiac or pulmonary insufficiency;
7. History of autoimmune diseases or immunodeficiency disorders;
8. Use of immunosuppressive drugs within the past year;
9. Distant metastasis to organs such as the abdominal cavity, pelvis, liver, or lungs;
10. Active bleeding;
11. Tumor involvement of adjacent structures such as the prostate or sacral organs, making the tumor unresectable;
12. Allergy to chemotherapeutic agents, immune checkpoint inhibitors, or cetuximab;
13. Psychiatric disorders or lack of capacity for civil conduct, unable to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete response rate | up to 2 months
  the incidence of no tumor residual after the treatment

IPD SHARING:
Plan to Share IPD: No